CLINICAL TRIAL: NCT01475409
Title: Dynamic Changes in IFN-gamma Plasma Levels Following Anti-TNF Treatment in Patients With Inflammatory Rheumatic Diseases Undergoing Serial QuantiFERON-TB Gold In-Tube Testing: a Prospective Study in a Low Tuberculosis Burden Country
Brief Title: A Study on Changes in IFN-gamma Levels Following Anti-TNF Treatment in Patients Undergoing Serial QuantiFERON-TB Gold In-Tube
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Rossana Scrivo, Principal Investigator, University of Roma La Sapienza
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: URomLS01
Record Dates: First submitted 2011-11-10; First posted 2011-11-21 (Estimated); Last update posted 2011-11-21 (Estimated); Status verified 2011-11

CONDITIONS: Inflammatory Rheumatic Diseases
Keywords: anti-TNF; tuberculosis; QuantiFERON-TB Gold In-Tube; tuberculin skin test; rheumatoid arthritis; spondyloarthritis
MeSH Terms: conditions — Tuberculosis; Arthritis, Rheumatoid; Spondylarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- QuantiFERON-TB Gold In-Tube (QFT-GIT) (Experimental): Patients were randomized to undergo, on the same day, tuberculin skin test (TST) and QFT-GIT by means of a randomization list to generate the order by which the 2 tests had to be executed. QFT-GIT was repeated after 3 and 6 months since TNF antagonist onset.
  Interventions: Biological: QuantiFERON-TB Gold In-Tube (QFT-GIT)

INTERVENTIONS:
Biological: QuantiFERON-TB Gold In-Tube (QFT-GIT) — Patients were randomized to undergo, on the same day, TST and QFT-GIT by means of a randomization list to generate the order by which the 2 tests had to be executed. QFT-GIT was repeated after 3 and 6 months since TNF antagonist onset

SUMMARY:
The screening for latent tuberculosis infection (LTBI) prior to the onset of anti-tumor necrosis factor therapy, as well as a watchful monitoring during the treatment, is strongly recommended. Tuberculin skin test (TST), universally used for this purpose, lacks sensitivity and specificity. The novel screening tools, including QuantiFERON-TB Gold In-Tube (QFT-GIT), have shown a higher specificity compared to TST, but their feasibility in the setting of immunosuppression remains unclear. Aims of this study were to investigate the performance of QFT-GIT and its agreement with TST in patients awaiting anti-tumor necrosis factor (TNF) therapy, and to evaluate the usefulness of serial QFT-GIT during the treatment with biologics to assess whether dynamic changes in interferon (IFN)-gamma levels may be helpful in identifying reactivation of LTBI or cases of newly acquired tuberculosis.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of inflammatory rheumatic diseases
* patients candidates to anti-TNF treatment

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2008-07; Primary Completion 2010-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in IFN-gamma plasma levels following serial QFT-GIT testing during the treatment with anti-TNF agents | From date of randomization (before anti-TNF treatment) until the date of repeated QFT-GIT testing (after 12 weeks and again after 24 weeks) for a total assessment of 7 months.
  QFT-GIT was performed at randomization (before commencement of anti-TNF treatment) and after 3 and 6 months since the beginning of biologicals.

SECONDARY OUTCOMES:
Performance of QFT-GIT and its agreement with TST in patients under consideration for anti-TNF agents | From date of randomization (before anti-TNF treatment) until the date of acquisition of QFT-GIT and TST results, for a total of 1 month.
  QFT-GIT and TST were performed at baseline, before the commencement of anti-TNF treatment.